CLINICAL TRIAL: NCT04439955
Title: A Phase 2a Placebo-controlled, Open-label, Single Center Study to Evaluate the Safety, Tolerability and Efficacy of Cannabidiol (CBD) as a Steroid-sparing Therapy in Chronic Spontaneous Urticaria (CSU) Patients
Brief Title: Study to Evaluate the Safety, Tolerability and Efficacy of Cannabidiol (CBD) as a Steroid-sparing Therapy in Chronic Spontaneous Urticaria (CSU) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stero Biotechs Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST-SCU-01
Record Dates: First submitted 2019-12-16; First posted 2020-06-19 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Intervention Model Description: Each patient will commence the study with a one month run-in period in which he/she will be administered individual with placebo (olive oil). At the end of the one month run-in period, all trial subjects will receive CBD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBD (Experimental): At the end of the one month run-in period, all trial subjects will continue on individual Standard of case plus increasing doses of CBD during the first six weeks of the study. Dosage of CBD will start at 25 mg twice a day and will be increased once every 14 days, if no side effects are observed, to 50 mg twice a day, 100 mg twice a day and finally to 150 mg twice a day CBD respectively. Treatment will be given with food. If the 300 mg CBD dose level is deemed safe for two weeks patients will continue receiving 300 mg CBD +for an additional follow-up period of three months
  Interventions: Drug: CBD

INTERVENTIONS:
Drug: CBD — 300 mg CBD

SUMMARY:
Each patient will commence the study with a one month run-in period in which he/she will be administered individual patient Standard of Care :anti-histamines and steroids as needed plus placebo (olive oil).

After the run-in period, doses of CBD will be incresed during the first six weeks of the study.

At the conclusion of the six weeks CBD dose escalation segment of the study, if the 300 mg CBD dose level is deemed safe for two weeks with standard of care doses of anti-histamines, patients will continue receiving 300 mg CBD with Anti-histamines as needed for an additional follow-up period of three month.

Each patient will serve as his/her own control.

DETAILED DESCRIPTION:
Each patient will commence the study with a one month run-in period in which he/she will be administered individual patient Standard of Care :anti-histamines and steroids as needed plus placebo (olive oil).

At the end of the one month run-in period, all trial subjects will continue on individual Standard of Care plus increasing doses of CBD during the first six weeks of the study. Dosage of CBD will start at 25 mg twice daily and will be increased once every 14 days, if no side effects are observed, to 50 mg twice a day, 100 mg twice a day and finally to 150 mg twice a day CBD respectively. Treatment will be given with food.

At the conclusion of the six weeks CBD dose escalation segment of the study, if the 300 mg CBD dose level is deemed safe for two weeks with standard of care doses of anti-histamines, patients will continue receiving 300 mg CBD with Anti-histamines as needed for an additional follow-up period of three months. In the case of flare, the patient will be treated with higher dose of Anti-histamines and Steroides if needed in addition to CBD. Once the flare has been brought under control, then another attempt will be made to discontinue the steroids and continue treating with CBD + Anti-histamines only. Each patient will serve as his/her own control.

Laboratory studies will be carried out at the beginning of the study (baseline), and then on a monthly basis until the end of the study.

Adverse events will be continuously assessed throughout the study

ELIGIBILITY:
Inclusion Criteria:

* Patients with active CSU for at least 4 months which was treated with anti-histamines as well as at least one course of steroids (ex. Prednisone)
* Age ≥18 years
* Patients will undergo an ECG and QT parameters will be measured for further analysis.
* Female subjects who are postmenopausal (absence of menses for ≥ 2 years confirmed by a follicle stimulating hormone test), or who are surgically sterilized may be enrolled. Similarly, women of childbearing potential who had a negative pregnancy test at screening, who are willing to use two medically acceptable methods of contraception for the duration of the study as well as for at least three months after cessation of CBD treatment and who are willing to undergo pregnancy testing according to the study protocol may be enrolled.
* Female subjects who are not breast-feeding and who have no intention to breast-feed during the term of the trial and for at least three months after cessation of CBD treatment may be enrolled.
* Subject able to provide written informed consent

Exclusion Criteria:

* Viral Hepatitis (HAV, HBV, HCV)
* HIV
* Serious psychiatric or psychological disorders
* Other chronic dermatological conditions under active treatment
* Active consumption of illicit drugs including cannabis or derivatives for at least three months prior to the study
* Patients with significant cardiac, respiratory or active malignance disease (except Basel Cell Carcinoma) comorbidities.
* Any uncontrolled infection at time of registration
* Renal comorbidity: eGFR < 30 mL/min/1.73m2 (note: CKD Grade 4 is defined as eGFR 15-29 mL/min/1.73 m2)
* Patient who is taking immunomodulatory medications for other indication
* Women of child-bearing potential who intend to become pregnant or who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Adverse Event reporting of up to 300 mg CBD/day | 6 month
  measured by Adverse Events significance of the difference in percent of subjects experienced any Adverse events, drug-related Adverse events and Serious Adverse events between the study groups
change in total steroid dose reporting | 6 month
  Total steroid dose needed to control flares during CBD administration period per patient versus the total steroid dose administered during the one month placebo run-in period
Number of days of flares | 6 month
  Total number of days of flares/month experienced per patient during CBD administration versus the total number of days of flares experienced during the one month placebo run-in period

SECONDARY OUTCOMES:
change in anti histamine use reporting | 6 month
  Percentage of patients who demonstrated a 50% reduction in anti-histamine use during the study
change in quality of life questionnaires | 6 month
  via UAS7, SF36, VAS, Cognitive QoL questionnaire, HDAS at baseline before initiation of CBD administration and at each clinical visit

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No